CLINICAL TRIAL: NCT03351088
Title: Outcomes of a Phase III Randomized Controlled Trial Comparing Preventive Versus Delayed Ligation of Dorsal Vascular Complex During Robot-assisted Radical Prostatectomy
Brief Title: Outcomes From a RCT Comparing Preventive Versus Delayed Ligation of DVC During Robot-assisted Radical Prostatectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Alessandro Antonelli, Dirigente medico, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DVC
Record Dates: First submitted 2017-11-19; First posted 2017-11-22 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preventive ligation (Other): Preventive ligation of DVC is done after the opening of endopelvic fascia and before bladder neck dissection. DVC is ligated at the level of the apex with a 8-fashion single stich (1-0 Monocryl® CT-1 stich) trying to preserve puboprostatic ligaments and the muscle fibres of the rabdosphincter. DVC is then dissected at the end of prostatectomy before the section of the urethra.
  Interventions: Procedure: DVC ligation
- Delayed ligation (Other): Delayed ligation is done after the section of the urethra and once the prostatectomy is completed with a single stich (3-0 Monocryl® UR-6).
  Interventions: Procedure: DVC ligation

INTERVENTIONS:
Procedure: DVC ligation — Ligation of the dorsal vascular complex during robot-assisted radical prostatectomy

SUMMARY:
Since its introduction, robot-assisted radical prostatectomy (RARP) have become the standard surgical approach for the treatment of prostate cancer in the United States and then in Europe. Continuous refinements of surgical technique has been described in order to maximise outcomes while minimizing morbidities.

The management of DVC is a crucial steps during RARP. It could be done prior or after its transection thanks to haemostatic effects of the pneumoperitoneum. This topic has been already investigated by some authors. However, no high quality evidence is available to opt in favour of either of the two approaches. Findings about estimated blood loss, positive surgical margins and urinary recovery differ among these studies and only one is a randomized controlled trial in a laparoscopic setting with a limited number of patients.

Therefore, our objective was to evaluate in a prospective randomised setting whether a delayed ligation of the dorsal vascular complex impacted on perioperative, functional and oncological outcomes as compared to preventive ligation during robot-assisted radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* male patients, aged 18-80 years
* patients willing and able to provide written informed consent
* voluntary partecipation
* clinical indication to robot-assisted radical prostatectomy

Exclusion Criteria:

* coagulation impairment at the time of surgery
* salvage radical prostatectomy

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Intraoperative estimated bool loss | intraoperative

SECONDARY OUTCOMES:
Transfusion rate | 30 days from surgery
Overall positive surgical marigins | intraoperative
Apical positive surgicals margins | intraoperative
1-month continence | 30 days from surgery
  0 or 1 security pad per day
1-month PSA | 30 days from surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Department of Urology, university Hospital Spedali Civili di Brescia, Brescia, Italy

IPD SHARING:
Plan to Share IPD: Undecided